CLINICAL TRIAL: NCT06804720
Title: Self-Compassion as a Well-Being Strategy Against Occupational Burnout in Dentistry: A Controlled Clinical Trial
Brief Title: Self-Compassion Against Burnout in Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cenk Haytac, Professor, Cukurova University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Cukurova University DHF-11
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Self Compassion; Mindfulness Meditation; Burn Out (Psychology)
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Self Compassion Training group) (Experimental)
  Interventions: Behavioral: Mindfulness based Self compassion
- Control group (No training) (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness based Self compassion — All participants in the test group completed the 8-week MBCL (Mindfulness-Based Compassionate Living) training, consisting of 2-hour sessions per week, in accordance with the MBCL training protocol. Training was conducted by one expert periodontist who is also an internationally certified MBCL instructor
  Arms: Test group (Self Compassion Training group)

SUMMARY:
Although studies have highlighted the relationship between stress-related psychopathological symptoms and changes in biochemical parameters, no study in dentistry has concurrently evaluated the association of stress and relaxation with biochemical markers and psychological parameters. Moreover, the impact of mindfulness-based self-compassion training programs on these variables has yet to be explored within this context. To enhance the well-being of dentists, an evaluation of a test group participating in an 8-week Mindfulness-Based Compassionate Living (MBCL) program was conducted. This assessment included daily cortisol curves, as well as salivary IL-6, IL-1β, and oxytocin levels. Additionally, empathy, burnout, self-compassion, depression, and mindfulness levels were measured before and after the training. In this study, the main hypothesis was that, compared to the control group, the test group would exhibit lower IL-1β, IL-6, and cortisol levels, along with higher oxytocin levels. Furthermore, as the secondary hypotheses was that the test group would demonstrate increased empathy, self-compassion, and mindfulness levels, accompanied by reductions in depression and burnout scores.

ELIGIBILITY:
Inclusion Criteria:

* dentists in their final year of specialty training at the Faculty of Dentistry,
* systemicaly healthy

Exclusion Criteria:

* individuals who received a diagnosis of mood disorders based on DSM-5 criteria following a standard diagnostic assessment conducted by psychiatrists from the Department of Psychiatry

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Scale | Baseline and after 8 weeks
  The 6 subscales that comprise the 26-item self-compassion scale are self-kindness, self-judgment , common humanity , isolation , mindfulness and over-identification Participants indicate their responses to each item using a 5-point scale ranging from 1 (Almost Never) to 5 (Almost Always). Higher score indicates greater self-compassion.

SECONDARY OUTCOMES:
Saliva Cortisol | Baseline and after 8 weeks
  Saliva sampling for the daily cortisol curve was scheduled for both the test and control groups. For the test group, samples were collected before the commencement of the MBCL (Mindfulness-Based Compassionate Living) training (T1) and after its completion (T2). For the control group, saliva collection was aligned with the same time periods with the test group. Samples were collected five times per day at specific time points: 30 minutes after waking, at 10:00 AM, 12:00 PM, 5:00 PM, and 10:00 PM (with group reminders provided at designated times). Salivary cortisol was estimated by solid phase enzyme-linked immunosorbent assay (ELISA) (DiaMetra, Boldon, UK) in ng/ml. The procedure was done as per the manufacturer guidelines on saliva samples.
Saliva IL 6 | Baseline and after 8 weeks
  IL-6 levels were measured in pg/ml using the commercial kit ELISA according to the instructions of the producer.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova UNiversity faculty of dentistry, Adana, Balcali, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No